CLINICAL TRIAL: NCT05140122
Title: The LEONIDaS(Long Term Exploration of Outcomes From New Interventions in Dravet Syndrome) Caregivers Study
Brief Title: LEONIDaS Caregivers Study
Acronym: LEONIDaS
Status: Withdrawn | Type: Observational
Why Stopped: Funder withdrew study before enrolment started..
Sponsor: University of Oxford (Other)
Collaborators: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R76178/RE001
Record Dates: First submitted 2021-10-22; First posted 2021-12-01 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Dravet Syndrome; Depression; Anxiety
MeSH Terms: conditions — Epilepsies, Myoclonic; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary caregivers of individuals with Dravet Syndrome
  Interventions: Drug: Multiple; Other: Multiple

INTERVENTIONS:
Drug: Multiple — We will collect information on all medications taken by the caregiver and the person they care for.
Other: Multiple — We will collect information on all forms of therapy or medical intervention taken by the caregiver and the person they care for.

SUMMARY:
Dravet syndrome is a rare form of severe epilepsy that begins in the first year of life and is associated with frequent and/or prolonged seizures. Individuals with Dravet Syndrome often experience a range of comorbidities, including behavioral and developmental delays, movement and balance issues, sleep difficulties, chronic infections, and growth and nutritional issues. Patients with Dravet syndrome are at high risk of death due to SUDEP (Sudden Unexpected Death in Epilepsy), prolonged seizures, seizure-related accidents, and infections.

Due to the severity of this condition, parents of children with Dravet syndrome are typically highly involved in their child's 24-hour care and this has a considerable impact on family life. Recent studies have highlighted the profound impact that such caregiving has on physical health, mental health, social function and financial resources. In particular, caregivers report high levels of stress and anxiety, fatigue, depression and social isolation. However, there is currently a lack of effective interventions to reduce the negative impact of caregiving on caregivers.

The aim of this study is to prospectively study carers of individuals with Dravet syndrome to identify pharmacological and psychological factors that are associated with increased or decreased vulnerability to stress, depression and anxiety. Using a naturalistic, observational design the investigators will assess a cohort of Dravet Syndrome carers every six months for 3 years in order to further characterise trajectories of caregiver burden and the factors that influence this, including factors related to the person with Dravet syndrome (e.g. age, seizure frequency/severity, treatment/medications, comorbidities) and factors related to the carer and family environment (e.g. social engagement/isolation, fatigue, finances, relationships). The investigators will use both standardized questionnaires and a neurocognitive task (Facial Expression Recognition Task) to assess vulnerability to anxiety and depression. The study will be conducted online.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Aged 18 years or above
* Primary caregiver of an individual with a medical history supporting a clinical diagnosis of Dravet syndrome
* Able to access the internet

Exclusion Criteria:

* Inability to provide informed written consent
* Another caregiver of the same individual with Dravet is already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of individuals with Dravet syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10-26 (Estimated); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression scores on the Hospital Anxiety and Depression Scale (HADS) | Follow up at three years
  Higher scores indicate higher symptom levels (worse outcome)
Anxiety and depression scores on the Hospital Anxiety and Depression Scale (HADS) | Follow up at two years
  Higher scores indicate higher symptom levels (worse outcome)
Anxiety and depression scores on the Hospital Anxiety and Depression Scale (HADS) | Follow up at one year
  Higher scores indicate higher symptom levels (worse outcome)
Caregiver stress scores on the UW Caregiver Stress Scale | Follow up at three years
  Higher scores indicate higher symptom levels (worse outcome)
Caregiver stress scores on the UW Caregiver Stress Scale | Follow up at two years
  Higher scores indicate higher symptom levels (worse outcome)
Caregiver stress scores on the UW Caregiver Stress Scale | Follow up at one year
  Higher scores indicate higher symptom levels (worse outcome)
Emotional processing biases on the Facial Expression Recognition Task (FERT) | Follow up at three years
Emotional processing biases on the Facial Expression Recognition Task (FERT) | Follow up at two years
Emotional processing biases on the Facial Expression Recognition Task (FERT) | Follow up at one year

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, PhD, Principal Investigator — University of Oxford